CLINICAL TRIAL: NCT06141031
Title: Phase I/IB Trial of Radiotherapy in Combination With TTI-101 in Borderline Resectable and Locally Advanced Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Tvardi Therapeutics, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 22-0734.cc; NCI-2023-10168 (Other: CTRP)
Record Dates: First submitted 2023-11-08; First posted 2023-11-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
Keywords: borderline resectable; locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — C188-9 compound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I (Experimental): During Phase 1, up to 2 dose levels of TTI-101 with SBRT will be tested using a 3 + 3 dose-escalation design to determine the RP2D. Up to 3 participants may be enrolled with either 0/3 or 1/3 DLT in order to more fully evaluate the safety and tolerability at a given dose level. Therefore, a minimum of 9 patients (3 at dose 0, and 6 at dose 1) and maximum 18 (6 patients at each dose level) will be enrolled in the phase 1.
  Interventions: Drug: TTI-101
- Phase II (Experimental): An additional 12 patients will be enrolled in phase 2 so that total of 18 patients are treated at RP2D in phase 2 (the 6 patients treated at RP2D in phase 1 will be rolled over to phase 2) of TTI-101 in combination with SBRT.
  Interventions: Drug: TTI-101

INTERVENTIONS:
Drug: TTI-101 — TTI-101 is an orally bioavailable, small-molecule inhibitor of Signal Transducer and Activator of Transcription 3 (STAT3), a transcription factor whose upregulation and activation governs many hallmarks of cancer, inflammation, and fibrosis.

SUMMARY:
To evaluate the safety and tolerability of TTI-101 given in combination with Stereotactic Body Radiation Therapy (SBRT) in borderline resectable and locally advanced pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed pancreatic adenocarcinoma with borderline resectable or locally advanced PDAC as defined by NCCN guidelines, with no expected arterial resection-reconstruction.
2. Borderline resectable patients only: Completion of inducation chemotherpy within 1-3 weeks of study treatment start. Patients that exceed this window should complete an additional cycle of induction chemotherapy prior to initiation of study treatment, per provider discretion.
3. Age ≥ 18 years at time of study entry.
4. Provision to sign and date the consent form.
5. Stated willingness to comply with all study procedures and be available for the duration of the study.
6. Ability to swallow tablets by mouth.
7. ECOG performance status ≤2 or KPS ≥60%
8. Absolute neutrophil count ≥ 1,000/mcL
9. Platelets ≥ 70,000/mcL
10. Hemoglobin ≥ 9 g/dL, patients may be transfused to meet this criterion
11. Serum albumin ≥ 2.8 g/dL
12. Total Bilirubin ≤ 2mg/dL
13. AST(SGOT)/ALT(SGPT)/ALP ≤ 3 x institutional upper limit of normal (IULN)
14. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL >40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 / 72 x serum creatinine (mg/dL)
15. INR ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
16. aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
17. Sexually active women of childbearing potential (defined in section 7.1) and men must agree to use at least 1 highly effective method of contraception (defined in section 7.1) from screening and for at least 30 days after administration of the last dose of the study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Exclusion Criteria:

1. Pregnant or breastfeeding. Patients must have a negative serum or urine pregnancy test within 5 days of study treatment.
2. Previous treatment of the current malignancy with a STAT inhibitor.
3. Herbal preparations are not allowed throughout the study. These herbal medications include but are not limited to St. John's wort, kava, ephedra (Ma Huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Participants should stop using herbal medications 7 days prior to the first dose of study treatment.

   a. Senna and flaxseed are permitted
4. Is not fully recovered from all COVID-19-related symptoms for 2 weeks prior to Cycle 1 Day 1, if previously tested positive for COVID-19.
5. Ongoing toxicity (except alopecia) due to a prior therapy, unless returned to baseline or Grade 1 or less.
6. Has had major surgery within 3 weeks prior to starting IP or has not recovered from major side effects due to surgery.
7. Significantly impaired cardiac function such as unstable angina pectoris, symptomatic congestive heart failure with New York Heart Association Class III or IV, myocardial infarction within the last 12 months prior to study entry; serious arrhythmia (including QTc prolongation of >470 ms and/or pacemaker) or prior diagnosis of congenital long QT syndrome.
8. Pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Participants with indwelling catheters for control of effusions or ascites are allowed.
9. History of cerebrovascular accident or stroke within the previous 2 years.
10. History of hepatic encephalopathy.
11. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected serum calcium >ULN).
12. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
13. History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition as TTI-101 (hydroxyl-naphthalene sulfonamides).
14. Known active metastases in the central nervous system (unless stable by brain imaging studies for at least 1 month without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants).
15. History of malabsorption, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the IP.
16. Participants with chronic HBV infection, unless screening viral load <500 IU/mL on stable doses of antiviral therapy. Note: Participants with chronic HCV infection are allowed to enroll into the study but do not have a defined maximum viral load requirement for study entry. Participants with both HBV and HCV infection are excluded unless they have negative HCV RNA.
17. History of malignancy other than PDAC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (eg, 5-year overall survival [OS] rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
18. Has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate participation in the clinical study, or compromise compliance with the protocol such as:

    * Chronic pancreatitis.
    * Active untreated or uncontrolled fungal, bacterial, or viral infections (including COVID-19), sepsis, etc.
    * Acute and chronic, active infectious disorders including viral and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy.
19. Prior treatment for pancreatic cancer in the past 2 years and outside of the induction chemotherapy received for the current diagnosis.
20. Measurable distant metastases on re-staging imaging post chemotherapy. tCurrently receiving any other investigational agents or has participated in a study of an investigational agent or using an investigational device overlapping with study treatments within 3-6 months preceding diagnosis at the discretion of the PI.
21. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to TTI-101.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by incidence of adverse events | 6 months
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes between baseline laboratory assessments | 2 years
  The PI will review and assess the changes in each participant's laboratory assessments to determine participants with abnormal laboratory values before, during, and after the delivery of SBRT in combination with TTI-101.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in electrocardiograms (ECGs) | 2 months
  The PI will review each participant's ECG before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patients blood pressure. | 6 months
  The PI will review each participant's blood pressure before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patient heart rate. | 6 months
  The PI will review each participant's heart rate before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patient SpO2. | 6 months
  The PI will review each participant's SpO2 before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patient weight. | 6 months
  The PI will review each participant's weight before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in abdominal distension of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in the abdominal distension by visual inspection and palpation on physical exam.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in tenderness to palpation on abdominal exam. of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in the tenderness to palpation on abdominal exam of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in ascites of each participant. | 6 months
  During the physical examination of each patient, the PI will assess any changes in ascites by a change in the level of dullness (shifting dullness) or demonstration of a transmitted fluid wave on physical exam.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in palpable gallbladder of each participant. | 6 months
  During the physical examination of each patient, the PI will assess any changes in the palpable gallbladder on inspiration in the region of the right mid-clavicular line and below the right costal margin.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in extremity edema of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in extremity edema of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in skin discoloration (jaundice) of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in skin discoloration (jaundice) of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in icteric sclera of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in icteric sclera of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in palmar erythema of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in palmar erythema of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in spider angioma of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in spider angioma of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in left supraclavicular lymphadenopathy (Virchow's node) of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in left supraclavicular lymphadenopathy (Virchow's node) of each participant.
Phase 1: Determine the safety of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in superficial thrombophlebitis (Trousseau's sign) of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in superficial thrombophlebitis (Trousseau's sign) of each participant.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by incidence of adverse events | 6 months
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes between baseline laboratory assessments | 2 years
  The PI will review and assess the changes in each participant's laboratory assessments to determine participants with abnormal laboratory values before, during, and after the delivery of SBRT in combination with TTI-101.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes between baseline ECGs | 2 months
  The PI will review each participant's ECG before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patients blood pressure. | 6 months
  The PI will review each participant's blood pressure before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patients heart rate. | 6 months
  The PI will review each participant's heart rate before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patients SpO2. | 6 months
  The PI will review each participant's SpO2 before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in patients weight. | 6 months
  The PI will review each participant's weight before and after the delivery of SBRT in combination with TTI-101 to determine any abnormal changes.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in abdominal distension of each participant. | 6 months
  During physical examination of each patient, the PI will assess any changes in the abdominal distension by visual inspection and palpation on physical exam.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in tenderness to palpation on abdominal exam of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the tenderness to palpation on abdominal exam of each participant.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in ascites of each participant. | 6 months
  During the physical examination of each patient, the PI will assess any changes in ascites by a change in the level of dullness (shifting dullness) or demonstration of a transmitted fluid wave on physical exam.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in palpable gallbladder of each participant. | 6 months
  During the physical examination of each patient, the PI will assess any changes in the palpable gallbladder on inspiration in the region of the right mid-clavicular line and below the right costal margin.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in extremity edema of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the extremity edema of each participant.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in skin discoloration (jaundice) of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the skin discoloration (jaundice) of each participant.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in the icteric sclera of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the icteric sclera of each participant.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in the palmar erythema of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the palmar erythema of each participant.
Phase 1: Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in the spider angioma of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the spider angioma of each participant.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in the left supraclavicular lymphadenopathy (Virchow's node) of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the left supraclavicular lymphadenopathy (Virchow's node) of each participant.
Phase 1: Determine the tolerability of delivering Stereotactic Body Radiation Therapy in combination with TTI-101 in borderline resectable pancreatic cancer by changes in the superficial thrombophlebitis (Trousseau's sign) of each participant. | 6 months
  During physical examination of each patient the PI will assess any changes in the left superficial thrombophlebitis (Trousseau's sign) of each participant.
Phase 2: To assess pathologic response rate (R0 resection) for those who revert to resectable status | 3 months
  To assess pathologic response rate (R0 resection) for those who revert to resectable status, compared to historical controls treated with SBRT alone

SECONDARY OUTCOMES:
Phase 1: Estimate Overall Response Rate by RECIST of the combination of TTI-101 + SBRT | 3 months
  To observe and record anti-tumor activity. Although the clinical benefit of this drug has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be monitored for response and survival outcomes in addition to safety and tolerability.
Phase 2: Determine the progression-free survival of the combination of TTI-101 plus stereotactic body radiation therapy | 2 years
  PFS will be compared to historical controls treated with the same regimen of hypofractionated radiotherapy alone
Phase 2: Determine the 2-year overall survival (OS) rate of patients treated with hypofractionated radiotherapy plus TTI-101 | 2 years
Phase 2: Evaluate the objective response rate (ORR, per RECIST 1.1) by imaging of patients treated with hypofractionated radiotherapy plus TTI-101 | 2 years
  ORR will be compared to historical controls treated with similar regimen on hypofractionated radiotherapy alone
Phase 2: Assess quality of life associated with treatment protocol using EORTC QLQ-C30 | 18 months
  Use a quality of life questionnaire at multiple time points using EORTC QLQ-C30. A higher score indicating a better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: David Binder, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No